CLINICAL TRIAL: NCT06013514
Title: A Prospective, Multi-center, Observational, Non Comparative, Post-marketing Surveillance Study to Obtain Clinical Outcome Data on the Nagor PERLE Range of Silicone Breast Implants When Used in Breast Implantation
Brief Title: Post-market Prospective Clinical Study of Nagor Perle Mammary Implants
Acronym: PERLE10PMCF
Status: Recruiting | Type: Observational
Sponsor: GC Aesthetics (Industry)
Responsible Party: Sponsor
Other Study IDs: DM6 640 0101
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Reconstruction; Breast Reconstruction Following Mastectomy; Breast Revision; Breast Augmentation; Breast Reconstruction With Silicone Implants; Breast Reconstruction After Mastectomy; Breast Reconstruction Surgery; Breast Implants
Keywords: prospective; observational; non-comparative; post-marketing study; PMCF; Perle; Nagor; GCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Smooth Silicone Breast Implant
  Interventions: Device: PERLE Sterile Smooth Opaque gel filled mammary implants

INTERVENTIONS:
Device: PERLE Sterile Smooth Opaque gel filled mammary implants — Sterile smooth opaque gel filled mammary implants will be implanted in adult women having breast surgery for either augmentation, reconstruction or revision surgery. Different ranges of implants will be used to suit patient needs

SUMMARY:
Patients can undergo breast implant surgery for multiple reasons; cosmetic and reconstructive being the primary indications. In order to confidently state safety and due to strict regulation on medical devices it is important to maintain a record of safety and performance with all medical implants.

This study is designed to collect data on a new generation of smooth mammary implants to assess the long term performance and safety data on this type of gel-filled mammary breast implant.

The two main complications of breast implants are capsular contracture and rupture; these complications can take years to develop. The study is designed to evaluate the occurrence of these two primary complication as well as other secondary complications over a period of 10 years. Patient follow up will be carried out pre-operatively and post operatively at 12 months and then 3, 5, 8 and 10 years thereafter.

The study will be carried out over 10 years to adequately assess complications which may only occur over the lifetime of the device such as systemic complications

ELIGIBILITY:
Inclusion Criteria:

1. Genetic female subjects aged ≥18 and ≤65
2. Subjects who underwent single or bilateral breast implantation with the study device for one of the following reasons:-

i) Primary breast reconstruction following mastectomy (both for one-stage or two-stage surgeries, including patients with previous radiotherapy and who have ADMs of animal origin (bovine, porcine)). ii) Primary breast augmentation (cosmetic surgery) with or without mastopexy iii) Breast revision surgery with or without mastopexy c) Subjects who have received a Nagor PERLE implant. d) Subjects who have provided informed consent and can adhere to the requirements of follow up appointments as per the study protocol.

Exclusion Criteria:

1. Subjects undergoing implant augmentation with a BMI > 30 and undergoing reconstruction with a BMI >32.
2. Subjects with autoimmune disease, lung fibrocystic disease, conditions that interfere with wound healing and blood clotting, a weakened immune system, reduced blood supply to the breast tissue or any other condition for which breast implants are contraindicated.
3. Subjects who have participated in a clinical study which involve chemical or drug study within 3 months prior to surgery, with the exception of subjects who are participating in breast cancer related clinical studies.
4. Subjects with insufficient tissue covering due to either radiation damage on the chest wall, tight thoracic skin grafts or radical resection of the pectoralis major muscle.
5. Subjects who have ADMs of synthetic origin.
6. Subjects who, in the Investigator's clinical opinion, have existing local or metastatic carcinoma of the breast that is unlikely to be fully excised at the time of insertion of the breast implant.
7. Subjects with known previous history of a sensitivity to silicone who, in the opinion of the Investigator, are unsuitable for surgery.
8. Subjects with an active infection who are unsuitable for surgery unless, in the opinion of the investigator, they are treated and cleared by the investigator.
9. Subjects with a history of abscesses anywhere in the body who, in the opinion of the Investigator, are unsuitable for surgery.
10. Subjects with a known history of compromised wound healing.
11. Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
12. Women who are pregnant and/or current breast feeders who do not stop breast feeding within 3 months of getting breast implants
13. Patients who have local recurrence or metastatic carcinoma at the time of insertion of breast implant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female 18-65 requiring breast surgery for iether augmentation, reconstruction or revision, meeting inclusion and non inclusion criteria
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2038-09 (Estimated); Study Completion 2038-09 (Estimated)

PRIMARY OUTCOMES:
Rate of capsular contracture (Baker grade III-IV) | 10 years post-surgery
Rate of implant rupture | 10 years post-surgery

SECONDARY OUTCOMES:
Rate of the secondary surgical procedures required for correction of complications | 10 years post-surgery
Rate and frequency of local complications associated with the use of Nagor gel-filled mammary implants | 10 years post-surgery
  * Capsular contracture of Baker Grade I-II
  * Haematoma
  * Rupture
  * Seroma
  * Severe and continuing pain
  * Post-operative infection
  * Explantation as a result of infection
  * Implant displacement/extrusion
  * Wrinkling/folds
  * Breast Implant Associate Anaplastic Large Cell Lymphoma
  * BII/Asia
  * Delayed or abnormal wound healing occurring within the first 3 months of surgery
  * Any other complications considered by the Investigator to be related to the device or surgical procedure
Patient satisfaction | 10 years post-surgery
  BREAST- Q method
rate and frequency of any adverse events | 10 years post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Manchester, Manchester, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: No